



## RESEARCH CONSENT FORM

| Name of Researcher(s) |
|---|
| Jayne Anderson (PhD student/ Chief Investigator), supervised by Professor Howard Hall, Dr. L. Samantha Yoward and Dr. Angela Green. |
| Title of study |
| Criterion validity of the Actigraph GT3X accelerometer in determination of body position and walking in hospital ward patients recovering from critical illness |
| Please read and complete this form carefully. If you would like to participate, please initial the box after each response and sign and date the declaration at the end of the consent form. |
| Patient ID Date of Birth |
| Please initial each respons |
| • I have had the study satisfactorily explained to me by the chief investigator and had the opportunity to read the information sheet dated (Version) |
| • I understand that the research will involve: |
| <ul> <li>Wearing two Actigraph GT3X accelerometers (activity<br/>monitors) secured with elastic belts, one on the mid - thigh<br/>and the other on the ankle of the same leg, each weighing 27g.</li> </ul> |
| O Completing a set of movements and body positions that I would usually perform during the day including lying on my bed, turning on my side, getting out of bed and getting back into bed, sitting in a chair, moving from my bed to my chair and taking a walk. I am free to perform these movements and body positions in any order I choose. I will be supervised by the chief investigator (Jayne Anderson, also a qualified physiotherapist) whilst I perform these movements, who will note each movement undertaken and the time when I start and finish them. |
| o Providing feedback of my view of how comfortable the accelerometers (activity monitors) were to wear. |
| • I understand that I am free to withdraw from this study without having to give any explanation. |
| • I understand that all information about me will be treated in strict confidence and I will not be identified in any presentations or written work, which will include a PhD thesis or journal publications. |

Version 1, Date: 1st April 2016



## Hull and East Yorkshire Hospitals

| <ul> <li>I understand that Jayne Anderson, the chief investigator will discuss the progress of the research with her supervision team named above.</li> <li>I understand that anonymous data collected during the study may be discussed with individuals from the PhD supervision team, regulatory authorities or the NHS Trust where it is relevant to my taking part in this research. I give my permission for these individuals to have access to these data.</li> <li>I give consent for my GP, or any other doctor treating me to be notified of my participation in the study.</li> </ul> | | | | | | |
|---|---|---|---|---|---|---|
| | | | | given a copy of th | is consent form for m | nis research study and have be<br>y own information, containing<br>ator and main supervisor. |
| | | | | Name of participant | Date | Signature |
| Name of person obtaining consent | Date | Signature | | | | |
| Preferred method of | contact if you would | l like to read a summary of th | ne study results: | | | |
| E-mail: | | | | | | |
| Telephone: | | | | | | |
| Postal address: | ••••• | •••••• | ••••• | | | |
| | ••••• | •••••• | ••••• | | | |

## **Chief Investigator Contact Details**

Jayne Anderson Grad. Dip. Phys. MCSP Lecturer Practitioner Physiotherapist/PhD Student Therapies Centre Hull Royal Infirmary Anlaby Road Hull HU3 2JZ

Tel: 01482 605293 (Direct) jayne.anderson@hey.nhs.uk

Version 1, Date: 1st April 2016

## **Main Supervisor Contact Details**

Professor Howard Hall
Chair in Sports Related Studies
De Grey Building,
York St John University
Lord Mayor's Walk
York
YO317EX
Tel: 01904 876302 (Direct)

Tel: 01904 876302 (Direct) h.hall@yorksj.ac.uk